CLINICAL TRIAL: NCT02976142
Title: Prospective Randomized Phase II Clinical Trial: the Efficacy of Surgical Treatment in Combinations With Intraperitoneal Immunotherapy and Systemic Chemotherapy in Patients With Gastric Cancer and Verified Free Cancer Cells
Brief Title: The Efficacy of Surgical Treatment After Neoadjuvant Chemotherapy Plus Intraperitoneal Immunotherapy Versus Chemotherapy Alone for Patients With Positive Wash Cytology Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKNC02/2016
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Gastric Cancer, Metastatic
Keywords: gastric cancer, metastatic; positive wash cytology; neoadjuvant intraperitoneal immunotherapy
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis

ARMS (2):
- neoadjuvant chemoimmunotherapy (Experimental): Patients with gastric cancer and verified free cancer cells who receive 1 course of intraperitoneal immunotherapy with interleykin-2 + 3 courses of systemic chemotherapy (Cisplatin + 5-FU). In case of downstaging (M1 -> M0) surgical treatment will be performed.
  Interventions: Procedure: neoadjuvant chemoimmunotherapy
- neoadjuvant chemotherapy (No Intervention): Patients with gastric cancer and verified free cancer cells who receive 3 courses of systemic chemotherapy (Cisplatin + 5-FU). In case of downstaging (M1 -> M0) surgical treatment will be performed.

INTERVENTIONS:
Procedure: neoadjuvant chemoimmunotherapy
  Arms: neoadjuvant chemoimmunotherapy

SUMMARY:
The purpose of this study is to determine whether intraperitoneal immunotherapy (with interleykin-2 - human cytokine reaction activator) with systemic chemotherapy will be more effective than systemic chemotherapy alone in patients with gastric cancer and verified free cancer cells in abdominal cavity in improving the long term outcomes and overall survival of further surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-2
* Histologically proven gastric cancer T2-3 N+, T4a with any N (0,+) with free cancer cells in the abdominal cavity and no macroscopic canceromathosis and no other distant metastases (TNM classification 7th edition)
* Histological forms: gastric adenocarcinoma and signet ring cancer
* Blood characteristics (creatinine <150 mg/l, total bilirubin < 50 mkmol/l, neutrophils < 1500/mkl, hemoglobin >90 g/l, thrombocytes > 100000/mkl)

Exclusion Criteria:

* Clinically apparent distant metastasis (besides free cancer cells)
* Synchronic or metachronic malignant tumors
* Previous systemic or surgical or combined therapy for gastric cancer
* Complications of gastric cancer (obstruction 0-1 GOOSS scale and/or gastric bleeding)
* Adhesions in abdominal cavity
* Gastrooesophageal junction cancer or gastric cancer with spreading on oesophagus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Overall 2-year survival | 2 years
  Overall 2-year survival for patients who received radical (R0) surgical treatment after downstaging (M1 -> M0; Cyt "+" -> Cyt "-") with initial free cancer cells in the abdominal cavity without macroscopic canceromathosis.

SECONDARY OUTCOMES:
Portability of the systemic therapy methods | 6,9,12,24 months
  Portability of the systemic therapy methods (intraperitoneal immunotherapy and systemic chemotherapy). Toxicity scale.
Mortality | 24 months
  Mortality related to intraperitoneal immunotherapy and systemic chemotherapy It is defined as the death within 24 months from the start of the treatment regardless of the reason.
Downstaging tumor | 2 years
  Number of patients that were downstaged (M1 -> M0; Cyt "+" -> Cyt "-") with initial free cancer cells in the abdominal cavity without macroscopic canceromathosis.
Morbidity | 30 days
  Number of postoperative morbidity and mortality in the early post-operative period (for patients who received radical (R0) surgical treatment after downstaging)
Quality of life | 6, 12, 18, 24 months
  Quality of life ECOG scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay Semenov, Principal Investigator — Moscow Clinical Scientific Center; Boris Pomortsev, Principal Investigator — Moscow Clinical Scientific Center